CLINICAL TRIAL: NCT00942630
Title: Percutaneous Cholangioscopy After Placement of a Percutaneous Transhepatic Biliary Drainage (PTBD) - a Prospective Study on Endoscopic Findings and Clinical Impact
Brief Title: Value of Percutaneous Cholangioscopy After Placement of a Percutaneous Transhepatic Biliary Drainage
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Tobias J. Weismueller, Dr. T. Weismüller, Hannover Medical School
Other Study IDs: MHH-ENDO-0709
Record Dates: First submitted 2009-07-20; First posted 2009-07-21 (Estimated); Last update posted 2011-10-10 (Estimated); Status verified 2011-10

CONDITIONS: Bile Duct Stricture Not Treatable by ERC
Keywords: percutaneous; transhepatic; biliary; drainage; cholangioscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In a prospective study the investigators perform repeated cholangioscopies in all patients that received percutaneous transhepatic biliary drainage (PTBD) for a variety of malignant and benign diseases. Endoscopic findings and their correlation with clinical features will be recorded prospectively. The impact on clinical decision will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

PTBD with at least 14 French in diameter

Exclusion Criteria:

missing informed consent

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients receiving a PTBD
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-12 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hannover Medical School, Hanover, Germany